CLINICAL TRIAL: NCT05964881
Title: PDS (Polydiaxonene Suture) Versus Prolene (Polypropylene Suture) as Suture Material for Vaginal Sacrospinous Hysteropexy - a Randomised Controlled Study
Brief Title: PDS Versus Prolene as Suture Material for Vaginal Sacrospinous Hysteropexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Greta L Carlin, Dr.med.univ, Dr. med. univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2079
Record Dates: First submitted 2023-06-20; First posted 2023-07-28 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Pelvic Organ Prolapse; Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDS - resorbable suture (Active Comparator): Operation through vaginal route, high posterior colpotomy is made towards the posterior cervix. Blunt preparation towards the right Spina ischiadica to visualise right sacrospinous ligament. PDS (0) sutures will be placed through the ligament (ca. 2 cm medial of the spina). This suture will then be placed through the posterior cervical wall, but not yet knotted. First, colpotomy will be closed via 2/0 vicryl, then pre-laid fixation sutures will be tied, whereby the portio will come to lie about 4-6 cm cranial of the level off the vulva towards the sacrospinous ligament.
  Interventions: Procedure: sacrospinous hysteropexy
- Prolene - non-resorbable sutures (Experimental): Operation through vaginal route, high posterior colpotomy is made towards the posterior cervix. Blunt preparation towards the right Spina ischiadica to visualise right sacrospinous ligament. Prolene (2-0) sutures will be placed through the ligament (ca. 2 cm medial of the spina). This suture will then be placed through the posterior cervical wall, but not yet knotted. First, colpotomy will be closed via 2/0 vicryl, then pre-laid fixation sutures will be tied, whereby the portio will come to lie about 4-6 cm cranial of the level off the vulva towards the sacrospinous ligament.
  Interventions: Procedure: sacrospinous hysteropexy

INTERVENTIONS:
Procedure: sacrospinous hysteropexy — sacrospinous hysteropexy

SUMMARY:
Introduction: Pelvic organ prolapse is a common gynecological disease, which about 50% of women develop in the course of their lives. There are many different options for surgical care, e.g. the uterus-preserving sacrospinal fixation (= sacrospinal hysteropexy = SSHP). This technique has been increasingly used in recent years. However, there is still no data on whether the fixation sutures should be performed with absorbable or non-absorbable threads. Internationally, both types of threads are routinely used and both types of threads are described in publications. So far, there is no comparative data on the effectiveness and subjective results. The aim of this study is to compare subjective symptom improvement Materials & Methods: This is a randomized, single-center superiority study. The sacrospinal fixation is performed according to a standardized method and two different types of threads (absorbable PDS sutures vs. non-absorbable Prolene sutures) are used for the fixation suture. Patients are randomized to either the absorbable PDS sutures group or the non-absorbable Prolene sutures group. The primary outcome of interest is the subjective symptom improvement 12 months after surgery (evaluated using the German version of the pelvic floor questionnaire). Secondary outcome variables are anatomical outcomes, condition-specific quality of life, and adverse events. 52 patients will be included in the study.

The results of the study will be published in peer-reviewed journals and the results will be presented at scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Anterior vaginal wall prolapse beyond the hymen (POP-Q-point Aa or Ba >0) with central defect
* Prolapse of the apical vaginal vault beyond the hymen (POP-Q point C >0) with central defect
* Symptoms of a vaginal bulge
* A primary reconstructive operation using sacrospinous hysteropexy is planned

Exclusion Criteria:

* Recurrent prolapse
* History of hysterectomy
* A primary reconstructive operation with mesh or obliterative surgery is planned
* An operation with hysterectomy is planned
* Known pelvic malignancy
* Known inflammatory disease
* Current systemic treatment with glucocorticoids or immunosuppressants
* The subject cannot or does not want to participate

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
German pelvic floor questionnaire (subjective symptom improvement) | 12 months post surgery
  subjective symptom improvement 12 months after surgery evaluated using the German version of the pelvic floor questionnaire, which consist of 4 domains and a total of 42 questions

SECONDARY OUTCOMES:
anatomical outcomes - POP-Q measurement | 12 months post surgery
  anatomical outcomes 12 months after surgery evaluated through POP-Q-system (standardised POP-Q scale ranging from 0-4; the higher the number the worse the prolapse)
anatomical outcomes - ultrasound imaging | 12 months post surgery
  anatomical outcomes 12 months after surgery evaluated through ultrasound (transvaginal ultrasound to measure size of uterus, length of cervix, perineal ultrasound for 3d imaging of perineal muscles)
German pelvic floor questionnaire (condition-specific quality of life) | 12 months post surgery
  condition-specific quality of life 12 months after surgery evaluated through validated german pelvic floor questionnaire (consisting of 4 domains and a total of 42 questions)
Clavien Dindo Scale for adverse events | 12 months post surgery
  assessment of adverse events during the first 12 months after surgery evaluated according to the Clavien Dindo scale from 1-5, with 5 consisting death)
Mini Nutritional Assessment | 12 months post surgery
  nutritional assessment 12 months after surgery (evaluated through Mini Nutritional Assessment (from 1-14 points: 12-14 points: normal nutrition, 8-11 points: at risk for malnutrition, 0-7 points: malnutrition)
Visual Analog Scale | 12 months post surgery
  pain assessment 12 months after surgery evaluated through Visual Analog Scale (VAS: pictograms of facial expression at different levels ranging from free of pain, to worst possible pain)
Numerical Rating Scale | 12 months post surgery
  pain assessment 12 months after surgery evaluated through Numeric Rating Scale (NRS: ranging from 0 (no pain) up to 10 (worst possible pain))
Patient Impression of Improvement Index | 12 months post surgery
  patient impression of improvment assessment 12 months after surgery evaluated through Patient Global Impression of Improvement Index (PGI-I: ranging from 1: very much better to 4: no change)

CONTACTS AND LOCATIONS:
Overall Officials: Greta L Carlin, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be public through upload on ClinicalTrials.gov Further information can be shared upon direct request from interested researchers
Supporting Information: Study Protocol, SAP
Time Frame: immediately
Access Criteria: Study Protocol and Statistical Analysis Plan will be accessible through ClinicalTrials.gov

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT05964881/Prot_SAP_000.pdf